CLINICAL TRIAL: NCT06912698
Title: A Phase III Randomized Controlled Non-Inferiority Clinical Trial Comparing Reduced-Dose Versus Standard-Dose Radiotherapy Based on Treatment Response in Early-Stage Nasopharyngeal Carcinoma
Brief Title: Reduced Dose Radiotherapy vs Standard Dose Radiotherapy for Early Stage Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hai-Qiang Mai,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-129
Record Dates: First submitted 2025-04-03; First posted 2025-04-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: radiotherapy; dose
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Reduced dose group (Experimental): Patients receive reduced dose radiotherapy.
  Interventions: Radiation: Reduced dose radiation
- Standard dose group (Active Comparator): Patients receive standard dose radiotherapy.
  Interventions: Radiation: Standard dose radiation

INTERVENTIONS:
Radiation: Reduced dose radiation — Reduced dose group would receive 61.48Gy radiation.
  Arms: Reduced dose group
Radiation: Standard dose radiation — Standard dose group would receive 69.96Gy radiation.
  Arms: Standard dose group

SUMMARY:
This study investigates whether administering reduced dose is non-inferior to standard dose radiotherapy in terms of 3-year locoregional relapse-free survival (LRRFS) rate for stage I nasopharyngeal carcinoma patients who are sensitive to radiotherapy.

DETAILED DESCRIPTION:
All the patients receive intensity-modulated radiotherapy. If patients receive CR and EBV DNA undetectable when completing 50.88Gy radiation, they will continue to receive radiotherapy until 61.48Gy, then the patients would be randomised assigned ( 1:1 ) to reduced dose group (observation) or standard dose group (continue to receive radiotherapy until 69.96Gy). Patients with stage IA will receive radiotherapy alone, and patients with stage IB will receive concurrent chemoradiotherapy. For patients with stage IB, those assigned to reduced dose group will receive a total of 2 cycles cisplatin concurrent chemotherapy, with 100mg/m2 per cycle; those assigned to standard dose group will receive a total of 3 cycles cisplatin concurrent chemotherapy, with 100mg/m2 per cycle. This study investigates whether administering reduced dose is non-inferior to standard dose radiotherapy in terms of 3-year locoregional relapse-free survival (LRRFS) rate for stage I nasopharyngeal carcinoma patients who are sensitive to radiotherapy. The primary endpoint is 3-year locoregional relapse-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, regardless of sex.
2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III, clinical stage I (according to the 9th American Joint Committee on Cancer[AJCC] edition).
3. Patients with CR according to RECIST and EBV DNA undetectable after received 50.88Gy radiation.
4. ECOG (Eastern Cooperative Oncology Group) score: 0-1.
5. Women in their reproductive years should ensure that they use contraception during the study period.
6. Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109 /L, platelet (PLT) ≥100×109 /L.
7. Liver function: Alanine transaminase(ALT), Aspartate aminotransferase(AST)< 1.5 times the upper limit of normal value (ULN), total bilirubin <1.5×ULN.
8. Renal function: serum creatinine <1.5×ULN or creatinine clearance rate≥60mL/min.
9. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I).
2. Patients with PR/SD/PD according to RECIST and/or EBV DNA detectable after received 50.88Gy radiation.
3. Receiving radiotherapy or chemotherapy or targeted therapy previously.
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
6. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
7. Severe, uncontrolled medical conditions and infections.
8. At the same time using other test drugs or in other clinical trials.
9. Refusal or inability to sign informed consent to participate in the trial.
10. Other treatment contraindications.
11. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2025-05-22 (Estimated); Primary Completion 2031-04-19 (Estimated); Study Completion 2033-03-19 (Estimated)

PRIMARY OUTCOMES:
Locoregional relapse-free survival | 3 year
  The time from randomization to either documented local and/or regional relapse or death from any cause,whichever occurred first.

SECONDARY OUTCOMES:
Progression-free survival | 3 year
  Time from randomisation to any documented local or regional relapse, distant metastasis, or death from any cause, whichever occurr first.
Overall survival | 3 year
  Time from randomisation to death from any cause or censored at the date of the last follow-up.
Distant metastasis-free survival | 3 year
  Time from randomistion to distant metastasis or death from any cause.
Incidence rate of adverse events (AEs) | 3 year
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Change of quality of life (QoL) score | 1 year
  QoL scores were assessed for each scale by using the European Organisation for Research and Treatment of Cancer (EORTC ) Quality of Life Questionnaire C30 (QLQ-C30) and EORTC QLQ-Head and Neck module (QLQ-H&N35) at 61.48Gy radiotherapy, at 1 month after radiotherapy, at 6 month after radiotherapy, and 12 month after radiotherapy.All of the scales and items ranged in score from 0 to 100. A high score for a functional or global QoL scale represents a relatively high/healthy level of functional or global QoL, whereas a high score for a symptom scale or item represents a high number of symptoms or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang MD, Dr., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mayr NA, Magnotta VA, Ehrhardt JC, Wheeler JA, Sorosky JI, Wen BC, Davis CS, Pelsang RE, Anderson B, Doornbos JF, Hussey DH, Yuh WT. Usefulness of tumor volumetry by magnetic resonance imaging in assessing response to radiation therapy in carcinoma of the uterine cervix. Int J Radiat Oncol Biol Phys. 1996 Jul 15;35(5):915-24. doi: 10.1016/0360-3016(96)00230-1. PMID 8751400
- [Background] Miao J, Di M, Chen B, Wang L, Cao Y, Xiao W, Wong KH, Huang L, Zhu M, Huang H, Huang S, Han F, Deng X, Xiang Y, Lv X, Xia W, Tan SH, Wee JTS, Guo X, Chua MLK, Zhao C. A Prospective 10-Year Observational Study of Reduction of Radiation Therapy Clinical Target Volume and Dose in Early-Stage Nasopharyngeal Carcinoma. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):672-682. doi: 10.1016/j.ijrobp.2020.03.029. Epub 2020 Apr 6. PMID 32272183
- [Background] Pan JJ, Mai HQ, Ng WT, Hu CS, Li JG, Chen XZ, Chow JCH, Wong E, Lee V, Ma LY, Guo QJ, Liu Q, Liu LZ, Xu TT, Gong XC, Qiang MY, Au KH, Liu TC, Chiang CL, Xiao YP, Lin SJ, Chen YB, Guo SS, Wong CHL, Tang LQ, Xu ZY, Jia YZ, Peng WS, Hu LP, Lu TZ, Jiang F, Cao CN, Xu W, Ma J, Blanchard P, Williams M, Glastonbury CM, King AD, Patel SG, Seethala RR, Colevas AD, Fan DM, Chua MLK, Huang SH, O'Sullivan B, Lydiatt W, Lee AWM. Ninth Version of the AJCC and UICC Nasopharyngeal Cancer TNM Staging Classification. JAMA Oncol. 2024 Oct 10;10(12):1627-35. doi: 10.1001/jamaoncol.2024.4354. Online ahead of print. PMID 39388190
- [Background] Rischin D, Corry J, Smith J, Stewart J, Hughes P, Peters L. Excellent disease control and survival in patients with advanced nasopharyngeal cancer treated with chemoradiation. J Clin Oncol. 2002 Apr 1;20(7):1845-52. doi: 10.1200/JCO.2002.07.011. PMID 11919243
- [Background] Songthong AP, Kannarunimit D, Chakkabat C, Lertbutsayanukul C. A randomized phase II/III study of adverse events between sequential (SEQ) versus simultaneous integrated boost (SIB) intensity modulated radiation therapy (IMRT) in nasopharyngeal carcinoma; preliminary result on acute adverse events. Radiat Oncol. 2015 Aug 8;10:166. doi: 10.1186/s13014-015-0472-y. PMID 26253488
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26253488/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11919243/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39388190/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32272183/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/8751400/